CLINICAL TRIAL: NCT07115316
Title: A RANDOMIZED, OPEN-LABEL TRIAL TO EVALUATE THE CLINICAL EFFECTIVENESS OF ECCENTRIC HAMSTRING CONTRACTIONS WITH PHYSIOTHERAPY TRAINING ON SPORTS PERFORMANCE AND QUALITY OF LIFE IN YOUNG MALE FOOTBALL PLAYERS WITH NON-CONTACT GRADE 1 ACL INJURY
Brief Title: EFFECTIVENESS OF ECCENTRIC HAMSTRING CONTRACTIONS WITH PHYSIOTHERAPY TRAINING ON SPORTS PERFORMANCE AND QUALITY OF LIFE IN YOUNG MALE FOOTBALL PLAYERS WITH NON-CONTACT GRADE 1 ACL INJURY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emirates Health Services (EHS) (Other Government)
Collaborators: Lincoln University College Malaysia (Other)
Responsible Party: Principal Investigator, Ajmal Sheriff, Physiotherapist, Emirates Health Services (EHS)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOHAP/DXB-REC/ J.F.M /No. 21/
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-08

CONDITIONS: Grade 1 Anterior Cruciate Ligament Injury
Keywords: Eccentric hamstring exercises, Grade 1 ACL Injury
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (conventional physiotherapy) (Active Comparator): Receives conventional physiotherapy alone
  1. Knee Straightening (Extension)
  2. Knee Bend (Flexion):
  3. Inner Range Quads
  4. Straight Leg Raise
  5. Lunge to Split Lunge
  6. Single Leg Sit to Stand
  7. Standing Hamstring Curls
  8. Double/Single Leg Bridge
  9. Side Lie Hip Abductions
  10. Crab Walks
  11. Forward Step Ups
  12. Calf Raises.
  13. Single Leg Balance
  14. Clock Face Mini Squat
  15. Arabesque Clock
  16. Two-Legged Jump / Single-Legged Hop
  Interventions: Other: Exercises
- Experimental Arm (Experimental): Receives both intervention exercises and conventional physiotherapy
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises — 1. Nordic hamstring curls
  2. Seated leg curls
  3. Prone leg curls
  4. Knee Straightening (Extension)
  5. Knee Bend (Flexion)
  6. Inner Range Quads
  7. Straight Leg Raise
  8. Lunge to Split Lunge
  9. Single Leg Sit to Stand
  10. Standing Hamstring Curls
  11. Double/Single Leg Bridge
  12. Side Lie Hip Abductions
  13. Crab Walks
  14. Forward Step Ups
  15. Calf Raises
  16. Single Leg Balance
  17. Clock Face Mini Squat
  18. Arabesque Clock
  19. Two-Legged Jump / Single-Legged Hop

SUMMARY:
The overall aim of the study is to evaluate the impact of eccentric hamstring contractions on sports performance in young male football players with non-contact grade 1 Anterior Cruciate Ligament injuries.

Treatment allocation will be assigned using an automated randomization process developed by an independent person who is not involved in the study. Computer-generated random numbers will be used for randomization into two groups.

Inclusion criteria Eligible patients with physician-diagnosed non-contact acute grade 1 ACL injury within the past 6 weeks will be invited from the selected clubs for participation in the trial. Participants who can perform full Range of Motion in the injured knee without pain will be included. Male football players between age 19-25 years old, currently playing in UAE, who speak English language and with physician-diagnosed non-contact grade 1 ACL injury will be included in the trial.

Exclusion Criteria

* Players with contact ACL injuries.
* Players with chronic grade 1 ACL Injuries.
* If pain and swelling are severe and occur within 24 hours after exercise, will be excluded from the study.
* Grade 2 and above ACL injuries.
* Female players.
* Players aged below 18 years or above 25 years.
* Players with a history of surgery on the same knee.
* Players with injuries to the menisci or other ligaments.
* Players who do not speak English.
* Players who refuse to provide written informed consent to participate in the trial.
* Players currently enrolled in other formal rehabilitation programs. There is no invasive procedure to be done. It focuses on strengthening the hamstrings muscle, specifically through eccentric contractions, which involve lengthening the muscle while it's under tension along with normal physiotherapy exercises.

The comparator group receives a variety of physiotherapy exercises aimed at improving strength, flexibility, and balance around the knee. For those patients who have mild pain or swelling will also be given TENS and Ultrasound.

DETAILED DESCRIPTION:
ACL injuries are prevalent in sports, particularly in activities that involve sudden stops, changes in direction, or direct impact on the knee. These injuries can have significant consequences, including pain, instability, and long-term joint damage(Montalvo et al., 2019). Understanding the mechanisms and risk factors for ACL injury is crucial for injury prevention and rehabilitation(Takahashi & Okuwaki, 2017). Eccentric contraction involves the elongation of a muscle while it is under tension. The hamstrings are a muscle group situated at the back of the thigh, comprising the biceps femoris, semitendinosus, and semimembranosus. The hamstrings play a crucial role in knee stability, particularly in preventing excessive anterior translation of the tibia relative to the femur, which is one of the mechanisms of ACL injury (Gronwald et al., 2022). Strengthening the hamstrings, especially through eccentric contractions, can enhance knee joint stability(Jones et al., 2019). Eccentric muscle contractions involve the lengthening of a muscle while it is contracting. These contractions are particularly effective in building strength and improving muscle function (Al Attar et al., 2017). Research suggests that eccentric hamstring strengthening exercises can enhance muscle activation, increase muscle strength, and improve neuromuscular control, all beneficial in ACL rehabilitation (Opar et al., 2012). Eccentric strengthening exercises for the hamstrings are commonly prescribed in rehabilitation programs for ACL injuries, because they provide dynamic stability to the knee joint (Lodge et al., 2019). ACL injury often occurs during dynamic movements such as cutting, pivoting, or landing from a jump. Biomechanical studies have identified specific movement patterns and muscle activation sequences associated with ACL injury risk (Buckthorpe et al., 2019).

Rehabilitation protocols for ACL reconstruction typically include strengthening exercises, neuromuscular training, proprioceptive exercises, and functional activities. Eccentric hamstring exercises are commonly incorporated into these programs to improve muscle strength, control, and proprioception around the knee joint(Vatovec et al., 2020).

Despite the widespread use of eccentric hamstring training in ACL rehabilitation after reconstruction, there may be gaps in our understanding of the effectiveness of eccentric hamstring contractions in ACL rehabilitation,for rehabilitation after ACLR, progressive eccentric cycle training was not more clinically effective than concentric training (Giovanni Milandri, Sudesh Sivarasu, 2021). Addressing these gaps can provide valuable insights for providing rehabilitation protocols and enhancing outcomes for individuals recovering from ACL injury.

Overall, the background of the study highlights the importance of understanding the relationship between eccentric hamstring contraction and ACL grade 1 injury rehabilitation. The study aims to provide insights into how eccentric hamstring contraction may influence ACL grade 1 injury rehabilitation.

4. THE OBJECTIVE OF THE STUDY

1. To assess the effectiveness of eccentric hamstring contractions on changes in sports performance, using various testing methods, in the intervention group.
2. To evaluate the impact of eccentric hamstring contractions on quality of life and psychological well-being in young male football players with non-contact grade 1 ACL injury.
3. To compare sports performance outcomes between the intervention and control groups in young male football players with non-contact grade 1 ACL injury.

The overall aim of the study is to evaluate the impact of eccentric hamstring contractions on sports performance in young male football players with non-contact grade 1 ACL injuries hamstring exercises on sports performance among young male football players with non-contact grade 1 ACL injury in UAE. The participants recruited in the study will be randomly assigned to one of two intervention groups: a control arm (usual physiotherapy exercise will be given) and, an intervention Arm (custom-tailored eccentric hamstring exercises along with physiotherapy will be given). We assumed no interaction between the treatment arms.

Operational Definitions

* ACL - The anterior cruciate ligament (ACL) is one of 2 cruciate ligaments that aids in stabilizing the knee joint. It is a strong band made of connective tissue and collagenous fibers that originate from the anteromedial aspect of the intercondylar region of the tibial plateau and extends posterolaterally to attach to the medial aspect of the lateral femoral condyle, where there are two important landmarks; The lateral intercondylar ridge which defines the anterior boundary of the ACL, and the bifurcate ridge which separates the 2 ACL bundles(Evans J, 2023).
* Eccentric hamstring exercises - An eccentric strengthening exercise program for the hamstring muscles that can be performed during training can help prevent hamstring injuries in soccer players(Schache A, 2012).
* Nordic hamstring curl training (NHCT), a type of training based on eccentric contractions aimed at increasing hamstring muscle strength and performed on flat ground without requiring special equipment, has been accepted as a popular training method(Al Attar, 2017).
* Running, one of the most basic human motions, is characterized by a typical cyclic motion and an airborne phase involving projection of the body. Sprint running is recognized as the fastest mode of unaided human locomotion (Michiyoshi Ae, 2017).

Pain Categories:

1. Mild: Pain intensity 1-3/10, occasional discomfort, no interference with daily tasks.
2. Moderate: Pain intensity 4-6/10, noticeable during activities, some difficulty with strenuous movements.
3. Severe: Pain intensity 7-10/10, significant pain at rest and with movement, difficulty with daily activities.

   * Swelling Categories:

1. Mild: Slight increase in size, no significant loss of motion, resolves with rest.

2. Moderate: Noticeable swelling, some difficulty with knee movement, lasts several hours or days.

3. Severe: Significant swelling, major restriction of movement, may require medical intervention.

ELIGIBILITY:
Inclusion Criteria:

* physician-diagnosed non-contact acute grade 1 ACL injury within the past 6 weeks will be invited from the selected clubs for participation in the trial. Participants who can perform full Range of Motion in the injured knee without pain will be included. Male football players between age 19-25 years old, currently playing in UAE, who speak English language and with physician-diagnosed non-contact grade 1 ACL injury will be included in the trial.

Exclusion Criteria:

* • Players with contact ACL injuries.

  * Players with chronic grade 1 ACL Injuries.
  * If pain and swelling are severe and occur within 24 hours after exercise, will be excluded from the study.
  * Grade 2 and above ACL injuries.
  * Female players.
  * Players aged below 18 years or above 25 years.
  * Players with a history of surgery on the same knee.
  * Players with injuries to the menisci or other ligaments.
  * Players who do not speak English.
  * Players who refuse to provide written informed consent to participate in the trial.
  * Players currently enrolled in other formal rehabilitation programs.

Ages: 19 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only male gender is involved in the study
Enrollment: 180 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Sargent vertical jump test | first intervention day and after 3 months
  The athlete warms up for 10 minutes. The athlete chalks the end of their fingertips. The athlete stands side onto the wall, keeping both feet remaining on the ground, reaches up as high as possible with one hand and marks the wall with the tips of the fingers (M1). From a static position, the athlete jumps as high as possible and marks the wall with the chalk on his fingers (M2).The therapist measures and records the distance between M1 and M2. The athlete repeats the test 3 times. The therapist calculates the average of the recorded distances and uses this value to assess the athlete's performance.

SECONDARY OUTCOMES:
• ACL Quality of Life (ACL-QOL) questionnaire | First day of intervention and after 3 months
  The ACL-QOL is a self-administered scale composed of 32 items divided into 5 domains: symptoms and physical complaints (5 items), work-related concerns (4 items), recreational activity and sport participation or competition Each domain has a proportional value according to the number of questions and is assessed with a 100-mm visual analog scale. A higher score indicates a better quality of life

OTHER OUTCOMES:
The Anterior Cruciate Ligament-Return to Sport after Injury scale (ACL-RSI). | First day of intervention and after 3 months
  The 12 questions on the ACL-RSI scale ask about the psychological effects of returning to sports. The ACL-RSI items are graded using either a VAS (visual analog scale) from 0 to 100 or an NRS (numeric rating scale) from 0 to 10. It has three domains: risk appraisal, confidence, and emotions. A total score between 0 and 100 is calculated by adding and averaging the scores for each item. Greater psychological preparation is indicated by higher scores
Psychological scoring using the Athletic Mental Energy Scale (AMES) questionnaire | First day of intervention and after 3 months
  The questionnaire comprises 18 interconnected questions. Respondents are required to select the most suitable level (ranging from completely so to totally inconsistent) from the 6 response options based on their own feelings. Each response option corresponds to a score (ranging from 6 to 1). The cumulative score serves as an indicator of participants' mental energy.

CONTACTS AND LOCATIONS:
Overall Officials: Anil John, PhD, Principal Investigator — Lincoln University College
Locations (1):
- Emirates Health services, Ras al-Khaimah, Emirate of Ras Al Khaimah, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
As per the informed consent

REFERENCES:
- [Background] Oliver GD, Dougherty CP. The razor curl: a functional approach to hamstring training. J Strength Cond Res. 2009 Mar;23(2):401-5. doi: 10.1519/JSC.0b013e31818f08d0. PMID 19204567
- [Background] Milandri G, Sivarasu S. A Randomized Controlled Trial of Eccentric Versus Concentric Cycling for Anterior Cruciate Ligament Reconstruction Rehabilitation. Am J Sports Med. 2021 Mar;49(3):626-636. doi: 10.1177/0363546520987566. Epub 2021 Feb 8. PMID 33555943
- [Background] Takahashi S, Okuwaki T. Epidemiological survey of anterior cruciate ligament injury in Japanese junior high school and high school athletes: cross-sectional study. Res Sports Med. 2017 Jul-Sep;25(3):266-276. doi: 10.1080/15438627.2017.1314290. Epub 2017 Apr 10. PMID 28391716